CLINICAL TRIAL: NCT02588794
Title: Cytokine Adsorption in Sepsis and Acute Kidney Injury
Acronym: CASAKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Guenther_Edenharter, Dr.med., Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 316/15 S
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Renal Insufficiency or Renal Failure &or End-stage Renal Disease
Keywords: sepsis, acute kidney injury , CytoSorb
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Sepsis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): Standart CVVHD plus CytoSorb 300 ml device (3804606CE01)
  Interventions: Device: CytoSorb 300 ml device (3804606CE01)
- control (No Intervention): Standart CVVHD

INTERVENTIONS:
Device: CytoSorb 300 ml device (3804606CE01) — additional cytokine adsorber
  Arms: intervention

SUMMARY:
Aim of the study is to reduce the incidence of RIFLE stadium L and E after acute kidney injury in patients with severe sepsis/septic shock

DETAILED DESCRIPTION:
Patient with proved severe sepsis/septic shock, treated in accordance to actual sepsis guidelines, who develope akute kidney injury (RIFLE I) or kidney failure (RIFLE F), were randomized in two groups.

One group is treated with CVVHD/ local citrat anticoagulation (standart clinical practice).

The other group ist treated with an additional cytokine adsorber ( 300ml CytoSorb device, 3804606CE01)

CytoSorb therapy is performed for 24h, then the adsorber is changed into a new device.

Cytosorb therapy is stopped, when Interleukin 6 leves drop below 1000 pg/ml in patient serum.

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis or septic shock according to ESICM guidelines not older than 24 h

Exclusion Criteria:

* preexisting renal disease KDIGO stadium 4 and 5

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
RIFLE stadium L or E after acute kidney injury related to sepsis | 3 months

SECONDARY OUTCOMES:
mortality | 3 months
length of renal replacement therapy | 3 months
SOFA score | 3 months
cumulative dose of vasopressor support | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kochs Eberhard, Chairman, Study Chair — Department of Anaesthsiology
Locations (1):
- Klinik für Anästhesiologie, München, Bavaria, Germany